CLINICAL TRIAL: NCT06770790
Title: Effect of Thoracic Epidural Anesthesia on Left Ventricular Functions: a Strain Echocardiography Study
Acronym: TEA-strain
Status: Not yet recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, asst.prof.dr, Aydin Adnan Menderes University
Other Study IDs: 199
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Thoracal Epidural Block; Echocardiography
Keywords: thoracic epidural anesthesia; left ventricle; strain echocardiography; cardiac function

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- thoracal epidural anesthesia: After appropriate local anesthesia, the patient will be placed in the epidural area while in a sitting position. The puncture will be performed between t6-t7 and t8-t9 with a midline approach with a "loss of resistance" specialist. The catheter is inserted into the epidural space 3-4 cm and the epidural lidocaine bolus (10 ml at 2% capacity) while the pain is in the supine region.
  Interventions: Other: strain echocardiography

INTERVENTIONS:
Other: strain echocardiography — HR, MAP, SBP, and DBP will be recorded at baseline and 15 minutes after ESP block. Cardiac output (CO) will be calculated using echocardiographic data on stroke volume (SV) (measured from the LV outflow tract) and multiplied by HR. Two transthoracic 2D echocardiographic examinations will be performed immediately before and 15 minutes after TEA. The examinations include apical four-, two-, and three-chamber projections, mitral and aortic Doppler flow velocities. Standard measurements of left ventricular systolic function include left ventricular volumes (indexed to body surface area, BSA), left ventricular ejection fraction (LVEF) according to the modified Simpson rule, time and velocity integral in the left ventricular outflow tract (TVI-LVOT), and stroke volume (SV) (= π x LVOT radius2 x TVI-LVOT). Stroke volume index (SVI) will be calculated as SV/BSA. Mitral and aortic Doppler flow profiles, left ventricular isovolumetric relaxation time, maximum flow velocity will be recorded for m

SUMMARY:
Post-thoracic surgery pain management thoracic epidural catheter is the most commonly used method.

Thoracic epidural anesthesia, in which cardiac sympathetic nerves (T1-T5) are involved in neural blockade, is the focus of our research. Many studies have shown a decrease in inotropic status (intrinsic function) after blockade of cardiac sympathetic innervation with thoracic epidural anesthesia (TEA).We want to examine the cardiac effects of TEA with strain echocardiography, which is an advanced echocardiography method. Therefore, we aimed to investigate the effect of TEA on left ventricular functions with strain echocardiography.

DETAILED DESCRIPTION:
The study was designed as an observational study. Our study will be conducted for 12 months after receiving ethical committee approval. 23 patients are planned to be included in the study. TTE will be performed when the patients arrive at the preoperative room for the operation. Then, thoracic epidural anesthesia will be performed. After the block, all usual medications, except ACE inhibitors, will be continued according to hospital protocol for 15 days of surgery. Patients will be given up to 2 mg midazolam and 7 ml/kg 0.5% isotonic 15 minutes before the epidural catheter is administered. A TTE will be performed before the epidural catheter is placed. After appropriate local anesthesia, the epidural catheter will be placed while the patient is in a sitting position. The puncture will be performed between t6-t7 and t8-t9 using the midline approach with the "loss of resistance" technique. The catheter will be inserted 3-4 cm into the epidural space and an epidural lidocaine bolus (10 ml at 2% concentration) will be administered while the patients are in the supine position. TTE will be performed again after 15 minutes. At these stages, hemodynamic values will also be recorded. We want to examine the cardiac effects of TEA with strain echocardiography, which is an advanced echocardiography method. Therefore, we aimed to investigate the effect of TEA on left ventricular functions with strain echocardiography.

ELIGIBILITY:
Inclusion Criteria:

Elective payment options ASA I-III Ages 18-75

Exclusion Criteria:

1. Refusal at enrollment
2. Request for withdrawal from the study
3. Inability to give informed consent
4. Emergency surgery
5. Bleeding diathesis
6. Presence of contraindications to the LA agents used in this study
7. Use of chronic opioids
8. Psychiatric disorders
9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will have a thoracic epidural catheter inserted for thoracic surgery and are between the ages of 18-75 and in the ASA1-3 group.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic assessment of left ventricular function | Left ventricular function will be assessed by echocardiography 15 minutes before and 15 minutes after high TEA.
  Description: Standard measurements of left ventricular systolic function include left ventricular volumes (indexed to body surface area, BSA), left ventricular ejection fraction (LVEF) according to the modified Simpson rule, time and velocity integral in the left ventricular outflow tract (TVI-LVOT), and stroke volume (SV) (= π x LVOT radius2 x TVI-LVOT). Stroke volume index (SVI) will be calculated as SV/BSA. Mitral and aortic Doppler flow profiles, left ventricular isovolumetric relaxation time, and maximum flow velocity measurements will be recorded. LV early (E-max) and late (A-max) diastolic filling will be assessed.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rex S, Missant C, Segers P, Wouters PF. Thoracic epidural anesthesia impairs the hemodynamic response to acute pulmonary hypertension by deteriorating right ventricular-pulmonary arterial coupling. Crit Care Med. 2007 Jan;35(1):222-9. doi: 10.1097/01.CCM.0000250357.35250.A2. PMID 17095942